CLINICAL TRIAL: NCT03515473
Title: Subjective and Objective Results With CI Electrode Types
Status: Completed | Type: Observational
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, László Rovó, Professor Head of Otorhinolaryngology Clinic, Szeged University
Other Study IDs: CI-001
Record Dates: First submitted 2018-01-15; First posted 2018-05-03 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Cochlear Implant
Keywords: cochlear implant; CI532; CI512; CI522; electrode array; perimodiolar; electrophysiology
MeSH Terms: interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- CI532: Patients with CI532 cochlear implant
  Interventions: Device: cochlear implant
- CI522: Patients with CI522 cochlear implant
  Interventions: Device: cochlear implant
- CI512: Patients with CI512 cochlear implant
  Interventions: Device: cochlear implant

INTERVENTIONS:
Device: cochlear implant — cochlear implant surgery

SUMMARY:
Background The authors' aim was to compare the influence of various electrode designs on selected objective and subjective clinical outcomes for cochlear implant recipients using the same model of receiver-stimulator, Cochlear™ Nucleus® Profile Series and sound processor.

Methods A multicenter study with subjects with profound sensorineural hearing loss, who were implanted and followed up in two tertiary centers. A total of 54 ears were implanted with Cochlear™ Nucleus® CI532, 51 with Cochlear™ Nucleus® CI522 and 54 with the Cochlear™ Nucleus® CI512. Implant loss and intraoperative electrophysiological tests (electrically evoked stapedial reflex threshold [ESRT], neural response telemetry threshold [T-NRT] and impedance), postoperative data (C-level, T-level, dynamic range, T-NRT and power consumption) and intracochlear position of the active electrode were analyzed with Nucleus Custom Sound 4.4 software.

ELIGIBILITY:
Inclusion Criteria:

* successful cochlear implantation with CI532 or CI512 or CI522
* gave informed consent

Exclusion Criteria:

* unsuccessful cochlear implantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects implanted with CI532 or CI512 or CI522 in Szeged and St. Pölten between the indicated time frames
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2017-06-04 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative measurements | 1 day
  Intraoperative impedance (kOhm) of the stimulating electrode with different types of cochlear implants.
Intraoperative measurements | 1 day
  Electrical stapedial reflex threshold (ESRT; current unit) with different types of cochlear implants
Intraoperative measurements | 1 day
  Neural response telemetry threshold (T-NRT; current unit) with different types of cochlear implants

SECONDARY OUTCOMES:
Postoperative measurements | 3 months
  Postoperative neural response telemetry threshold (T-NRT; current unit) with different types of cochlear implants
Postoperative measurements | 3 months
  Postoperative comfort level (C-level; current unit) with different types of cochlear implants
Postoperative measurements | 3 months
  Power consumption of different types of cochlear implants

CONTACTS AND LOCATIONS:
Locations (1):
- Universitiy of Szeged, Department of Otorhinolaryngology, Head and Neck Surgery, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No